CLINICAL TRIAL: NCT00424606
Title: A Multicenter Randomized Phase III Study of Adjuvant Treatment With Epirubicin Followed by Docetaxel (E/T) Versus Epirubicin and Docetaxel Combination (ET) in High Risk Lymph Node Negative Breast Cancer Patients
Brief Title: Epirubicin and Docetaxel Combination (ET) or Epirubicin Followed by Docetaxel (E/T) for Node Negative (N0) High Risk Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/01.04
Record Dates: First submitted 2007-01-18; First posted 2007-01-19 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer
Keywords: High risk node negative
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Docetaxel; Drug: Epirubicin
- 2 (Experimental)
  Interventions: Drug: Epirubicin; Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Docetaxel at the dose of 75 mg/m2 intravenously (IV) every 3 weeks for 4 consecutive cycles
  Other Names: Taxotere
  Arms: 1
Drug: Epirubicin — Epirubicin at the dose of 90 mg/m2 IV every 3 weeks for 4 consecutive cycles
  Other Names: Farmorubicin
  Arms: 1
Drug: Epirubicin — Epirubicin at the dose of 75 mg/m2 IV every 3 weeks for 6 consecutive cycles
  Other Names: Farmorubicin
  Arms: 2
Drug: Docetaxel — Docetaxel at the dose of 75 mg/m2 IV every 3 weeks for 6 consecutive cycles
  Other Names: Taxotere
  Arms: 2

SUMMARY:
The combination of taxanes, and especially docetaxel, with an anthracycline seems to be an important part of the chemotherapy regimens used in the adjuvant setting of patients with early-stage node-positive breast cancer patients. Whether sequential or concurrent administration of these drugs is preferable is not yet known, especially in patients with node-negative high risk tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast adenocarcinoma.
* Within 20-45 days after the surgical excision of the primary tumor with tumor-free operation margins; at least 10 axillary lymph nodes have to be removed.
* Absence of lymph node involvement after eclosion and hormone (E&H) staining and light microscopy evaluation.
* Premenopausal or postmenopausal women with at least one of the following tumor characteristics is required in order to characterize the tumor as high risk:

  * Estrogen receptor (ER) (-) and progesterone receptor (PR)(-);
  * Ki-67 + > 30%; Grade III; HER2 (3+) (after an amendment on 15.05.2008 women with HER2 (3+) were not included); Perineural infiltration or presence of tumor emboli in blood or lymph vessels.
* Postmenopausal women with tumors 1-2 cm are eligible if the tumor has at least 2 of the above mentioned high risk criteria.
* Premenopausal and postmenopausal women with tumors measuring > 2 cm are eligible irrespectively of the expression of the above adverse prognostic tumor criteria.
* Absence of any clinical or radiological evidence of local or metastatic disease.
* Age > 18 years.
* Performance status (WHO) < 3.
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9 gr/mm^3).
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2 mg/dl).
* Adequate cardiac function (LVEF > 50%).
* Negative pregnancy test.
* Informed consent.

Exclusion Criteria:

* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer.
* Other concurrent uncontrolled illness that could affect compliance with the study.
* Psychiatric illness or social situation that would preclude study compliance.
* Pregnant or nursing women.
* History of allergic reaction attributed to docetaxel.
* Other concurrent investigational agents.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2001-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Disease-free interval between the two treatment arms | Five years

SECONDARY OUTCOMES:
Comparison of overall survival and safety between the two treatment arms | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Mavrudis, MD, Principal Investigator — University Hospital of Heraklion Dept. of Medical Oncology
Locations (12):
- Greece (12):
  - University Hospital of Heraklion, Heraklion, Crete
  - University Hospital of Alexandroupolis Dept. of Medical Oncology, Alexandroupoli
  - "Agios Savvas" Anticancer Hospital of Athens, Athens
  - "IASO" General Hospital of Athens, Athens
  - "Laikon" General Hospital, Athens
  - "Marika Iliadis" Hospital of Athens, Athens
  - "Metaxa's" Anticancer Hospital of Pireas, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - State General Hospital of Larissa, Larissa
  - "AXEPA" General Hospital of Thessaloniki, Thessaloniki
  - "Theagenion" Anticancer Hospital of Thessaloniki, Thessaloniki